CLINICAL TRIAL: NCT00006358
Title: Phase II Evaluation of Temozolomide (SCH52365) and Thalidomide for the Treatment of Recurrent and Progressive Glioblastoma Multiforme
Brief Title: Temozolomide Plus Thalidomide in Treating Patients With Recurrent or Progressive Brain Tumor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Treatment
Other Study IDs: NABTC-9904; CDR0000068227 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2000-10-04; First posted 2004-05-26 (Estimated); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: recurrent adult brain tumor; adult glioblastoma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms; Glioblastoma; Gliosarcoma | interventions — Temozolomide; Thalidomide

INTERVENTIONS:
Drug: temozolomide
Drug: thalidomide

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Thalidomide may stop the growth of cancer by stopping blood flow to the tumor.

PURPOSE: Phase II trial to study the effectiveness of combining temozolomide and thalidomide in treating patients who have recurrent or progressive brain tumor.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the efficacy of temozolomide and thalidomide in patients with recurrent or progressive supratentorial glioblastoma multiforme or gliosarcoma. II. Determine the toxicity of this regimen in these patients.

OUTLINE: This is a multicenter study. Patients receive oral temozolomide once daily on days 1-5 and oral thalidomide daily on days 1-28. Treatment repeats every 28 days for a maximum of 24 courses in the absence of disease progression or unacceptable toxicity. Patients are followed at 1 month and then for survival.

PROJECTED ACCRUAL: A total of 40 patients will be accrued for this study within 4-5 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed supratentorial glioblastoma multiforme or gliosarcoma Must have evidence of tumor recurrence or progression by MRI scan after failing prior radiotherapy Bidimensionally measurable enhancing residual disease on MRI or CT scan Prior recent resection of recurrent or progressive tumor allowed if all of the following conditions apply: Recovered from surgery Residual evaluable disease present that is not artifactual postsurgical enhancement Baseline MRI or CT scan is performed within 14 days prior to study and while on a steroid dose that has been stable for at least 5-7 days

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 60-100% Life expectancy: At least 8 weeks Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: SGPT less than 2 times normal Alkaline phosphatase less than 2 times normal Bilirubin less than 1.5 mg/dL Renal: BUN or creatinine less than 1.5 times normal Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use one highly effective method of contraception, AND one additional effective method of contraception for at least 4 weeks before, during, and for 8 weeks after study No peripheral neuropathy greater than grade 1 No active infection No other illness that would obscure toxicity or alter drug metabolism No other concurrent serious medical illness No other prior cancer within the past 3 years except nonmelanoma skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior thalidomide No other concurrent biologic therapy for cancer Chemotherapy: No more than 1 prior chemotherapy regimen At least 3 weeks since prior chemotherapy (2 weeks for vincristine and 6 weeks for nitrosoureas) No other concurrent chemotherapy for cancer Endocrine therapy: See Disease Characteristics No concurrent endocrine therapy for cancer Radiotherapy: See Disease Characteristics No concurrent radiotherapy for cancer Surgery: See Disease Characteristics No concurrent surgery for cancer Other: Recovered from prior therapy No other concurrent investigational drugs for cancer

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2000-06-13 (Actual); Primary Completion 2003-01-23 (Actual); Study Completion 2006-07-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Morris D. Groves, MD, JD, Study Chair — M.D. Anderson Cancer Center
Locations (11):
- United States (11):
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - Neuro-Oncology Branch, Bethesda, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin

REFERENCES:
- [Result] Groves MD, Puduvalli VK, Chang SM, Conrad CA, Gilbert MR, Tremont-Lukats IW, Liu TJ, Peterson P, Schiff D, Cloughesy TF, Wen PY, Greenberg H, Abrey LE, DeAngelis LM, Hess KR, Lamborn KR, Prados MD, Yung WK. A North American brain tumor consortium (NABTC 99-04) phase II trial of temozolomide plus thalidomide for recurrent glioblastoma multiforme. J Neurooncol. 2007 Feb;81(3):271-7. doi: 10.1007/s11060-006-9225-y. Epub 2006 Sep 22. PMID 17031561